CLINICAL TRIAL: NCT03880942
Title: The Effect of Reading an Informative Story Book on Preoperative Anxiety
Brief Title: The Effect of Reading Book on Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, gözde bumin aydın, associate professor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 55/13
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Preoperative Anxiety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informative Story Book (Active Comparator): Patients will be given a colorful story book that tells the hospital and operation procedure named 'Elif Ameliyat Oluyor'(Elif is undergoing surgery) and will be asked to read the book with children at least once before the operation.
  Interventions: Other: Informative story book
- Non Informative Story Book (Placebo Comparator): Patients will be given a non-medical colorful story book called 'Çiftlik Öyküleri-Kamp' (Farm Stories-Camp) and will be asked to read the book with children at least once before the operation.
  Interventions: Other: Non Informative Story Book

INTERVENTIONS:
Other: Informative story book — Patients will be given a colorful story book that tells the hospital and operation procedure named 'Elif Ameliyat Oluyor'(Elif is undergoing surgery) and will be asked to read the book with children at least once before the operation.
  Other Names: Elif Ameliyat Oluyor
  Arms: Informative Story Book
Other: Non Informative Story Book — Patients will be given a non-medical colorful story book called 'Çiftlik Öyküleri-Kamp' (Farm Stories-Camp) and will be asked to read the book with children at least once before the operation.
  Other Names: Çiftlik Öyküleri-Kamp
  Arms: Non Informative Story Book

SUMMARY:
Observe the effects of reading an informative story book on preoperative anxiety and maternal anxiety

DETAILED DESCRIPTION:
Observe the effects of reading an informative story book at preoperative period on preoperative anxiety by m-YPAS in the holding area and on maternal anxiety by STAI in the holding area.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Elective surgery

Exclusion Criteria:

* Chronic diseases
* Development disability
* Prematurity
* Neurological diseases
* Psychoactive medication use
* Hearing/visual impairment
* History of surgery

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
preoperative anxiety | Preoperative anxiety will be evaluated at two times. At the preoperative holding area before given premedication and while entering to the operating room.
  Preoperative anxiety will be evaluated by mYPAS (modified Yale Preoperative Anxiety Scale) The mYPAS consists of 22 items in five categories (activity, emotional expressivity, state of arousal, vocalization and use of parents). The highest behavioral level observed in each of the five mYPAS categories is the score for that category. Partial weights were calculated and then added to a total score that ranged from 0 to 100. Cut off points were set to classify: a score of 23.4 to 30 for no anxiety, any score greater than 30 for anxiety.
  Preoperative anxiety at preoperative waiting room and at operation room will be evaluated.

SECONDARY OUTCOMES:
maternal anxiety | It will be evaluated once. At the preoperative holding area while waiting for operation with their child.
  Maternal state anxiety will be evaluated by STAI-FORM TX1 questionnaire at preoperative waiting room.
  The STAI TX1 is an internationally well accepted measure and has been used in a range of comparable studies for assessing the level of parents'anxiety. Raw scores on each subscale range between 20 and 80, with higher scores reflecting higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- DiskapiYBERH, Ankara, Turkey (Türkiye)